CLINICAL TRIAL: NCT05767658
Title: Support Via Online Social Networks to Promote Safe Infant Care Practices Toward Reducing Racial Disparities in Infant Mortality
Brief Title: Support Via Online Social Networks to Promote Safe Infant Care Practices
Acronym: SUPERSONIC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: Boston University (Other); Washington University School of Medicine (Other); Boston Medical Center (Other); University of Kentucky (Other); National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Rachel Moon, MD, Professor, Department of Pediatrics, University of Virginia
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: H-43455; 5R01MD007702-07 (NIH)
Record Dates: First submitted 2023-03-02; First posted 2023-03-14 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Breastfeeding; Infant Death; Sudden Infant Death Syndrome Without Mention of Autopsy
Keywords: Safe Sleep; Breastfeeding; Social Media
MeSH Terms: conditions — Breast Feeding; Infant Death | interventions — Lactation

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Safe Sleep (Experimental): Participants will be part of a private Facebook group from approximately 32 weeks gestation to 6 months postpartum. The Facebook group will provide a) evidence-based education through videos and other multi-media supporting best practices for infant safe sleep and b) an online community and social network of other pregnant WIC clients and new parents
  Interventions: Behavioral: Safe Sleep
- Breastfeeding (Experimental): Participants will be part of a private Facebook group from approximately 32 weeks gestation to 6 months postpartum. The Facebook group will provide a) evidence-based education through videos and other multi-media supporting best practices for breastfeeding and b) an online community and social network of other pregnant WIC clients and new parents
  Interventions: Behavioral: Breastfeeding
- Safe Sleep and Breastfeeding (Experimental): Participants will be part of a private Facebook group from approximately 32 weeks gestation to 6 months postpartum. The Facebook group will provide a) evidence-based education through videos and other multi-media supporting best practices for infant safe sleep and breastfeeding, and b) an online community and social network of other pregnant WIC clients and new parents
  Interventions: Behavioral: Safe Sleep; Behavioral: Breastfeeding
- Early Brain Development and Parent -Child Relationships (Active Comparator): Participants will be part of a private Facebook group from approximately 32 weeks gestation to 6 months postpartum. The Facebook group will provide a) evidence-based education through videos and other multi-media supporting best practices for early brain development and parent-child interactions (control intervention) and b) an online community and social network of other pregnant WIC clients and new parents.
  Interventions: Behavioral: Early Brain Development and Parent-Child Relationships

INTERVENTIONS:
Behavioral: Safe Sleep — Participants will be part of a private Facebook group from approximately 32 weeks gestation to 6 months postpartum. The Facebook group will provide a) evidence-based education through videos and other multi-media supporting best practices for infant safe sleep and b) an online community and social network of other pregnant WIC clients and new parents.
  Arms: Safe Sleep; Safe Sleep and Breastfeeding
Behavioral: Breastfeeding — Participants will be part of a private Facebook group from approximately 32 weeks gestation to 6 months postpartum. The Facebook group will provide a) evidence-based education through videos and other multi-media supporting best practices for breastfeeding and b) an online community and social network of other pregnant WIC clients and new parents.
  Arms: Breastfeeding; Safe Sleep and Breastfeeding
Behavioral: Early Brain Development and Parent-Child Relationships — Participants will be part of a private Facebook group from approximately 32 weeks gestation to 6 months postpartum. The Facebook group will provide a) evidence-based education through videos and other multi-media supporting best practices for early brain development and parent-child interactions (control intervention) and b) an online community and social network of other pregnant WIC clients and new parents.
  Arms: Early Brain Development and Parent -Child Relationships

SUMMARY:
This study aims to improve adherence to American Academy of Pediatrics safe sleep (SS) recommendations and improve rates of initiation and duration of partial and exclusive breastfeeding (BF); and reduce Black/White disparities in these practices through the use of private Facebook groups providing a) evidence-based education through videos and other multi-media supporting best practices and b) an online community and social network of other pregnant WIC clients and new parents.

ELIGIBILITY:
Inclusion Criteria:

* Currently enrolled in WIC, or it not, then have either Medicaid or no health insurance
* Must be English speaking
* Must be pregnant and less than 30 weeks gestation
* Must live in the United States
* Must have regular access to Facebook and short message service (SMS) texting (mobile phone)

Exclusion Criteria:

* Not planning to live in same home as infant after birth.
* Prenatal diagnosis expected to impact on infant care practices in a manner not compatible with study goals, including contraindications to feeding any breastmilk or supine infant sleep positioning.
* Known or reported mental health or other issues that would preclude custody of the infant or being able to participate in the informed consent process.
* Meets the definition of a minor according to applicable state law.
* Participants who consent to participation in the study, must complete the Agile Onboarding process before they reach 30+0 weeks gestation.
* Currently or previously received a TodaysBaby educational program (randomized to a TodaysBaby program through either the SMARTER, or SUPERSONIC study), either in their current or a previous pregnancy.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3000 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Exclusive infant supine sleep position in the previous two weeks | Between 2 and 6 months
  An investigator-developed maternal survey will be used to assess infant's usual sleep position during the previous two weeks with categorical responses of back, stomach, side, and other, with the proportion of infants using exclusive supine sleep position as the primary outcome measure.
Infant sleep location (exclusive room sharing without bed sharing) in the previous two weeks | Between 2 and 6 months
  An investigator-developed maternal survey will be used to assess the infant's usual sleep location during the previous two weeks with categorical responses of room sharing without bed sharing, room sharing with bed sharing, no room sharing and no bed sharing, with the proportion of infants exclusively room sharing without bed sharing as the primary outcome measure.
Soft bedding use in the previous two weeks | Between 2 and 6 months
  An investigator-developed maternal survey will be used to assess soft bedding placed in and around the infant (while sleeping) during the previous two weeks with categorical responses of Yes or No.
Breastmilk feeding in the previous two weeks | Between 2 and 6 months
  An investigator-developed maternal survey will be used to assess whether the infant was breast fed during the previous two weeks with categorical responses of exclusively breast fed, partially breast fed, or not breast fed.

SECONDARY OUTCOMES:
Usual infant sleep position in the previous two weeks | Between 2 and 6 months
  An investigator-developed maternal survey will be used to assess infant's usual sleep position during the previous two weeks with categorical responses of back, stomach, side, and other.
. Usual infant sleep location in the previous two weeks | Between 2 and 6 months
  An investigator-developed maternal survey will be used to assess the infant's usual sleep location during the previous two weeks with categorical responses of room sharing without bed sharing, room sharing with bed sharing, no room sharing and no bed sharing.
Pacifier use in the previous two weeks | Between 2 and 6 months
  An investigator-developed maternal survey will be used to assess the infant's pacifier use during the previous two weeks with categorical responses of Yes or No.

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Y Moon, MD, Principal Investigator — University of Virginia School of Medicine
Locations (1):
- Boston University Medical Campus, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No